CLINICAL TRIAL: NCT02315417
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Gevokizumab in Treating Active Ulcers of Pyoderma Gangrenosum
Brief Title: An Efficacy and Safety Study of Gevokizumab in Treating Active Ulcers of Pyoderma Gangrenosum
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X052172; NCT02366260 (obsolete NCT alias)
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Pyoderma Gangrenosum
Keywords: Pyoderma Gangrenosum; Classic Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- gevokizumab (Experimental): Solution for subcutaneous injection (Part 1, Group B)
  Interventions: Drug: gevokizumab
- Placebo (Placebo Comparator): Solution for subcutaneous injection (Part 1, Group A)
  Interventions: Drug: Placebo
- gevokizumab open-label (Experimental): Solution for subcutaneous injection (Part 2, Open-label)
  Interventions: Drug: gevokizumab open-label

INTERVENTIONS:
Drug: gevokizumab
  Arms: gevokizumab
Drug: Placebo
  Arms: Placebo
Drug: gevokizumab open-label
  Arms: gevokizumab open-label

SUMMARY:
The study will evaluate the efficacy and safety of gevokizumab in treating active ulcers of pyoderma gangrenosum (PG).

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of classic pyoderma gangrenosum
* An active pyoderma gangrenosum ulcer
* Contraceptive measures adequate to prevent pregnancy during the study

Exclusion Criteria:

* Clinical evidence of acutely infected pyoderma gangrenosum
* History of allergic or anaphylactic reactions to monoclonal antibodies
* History of recurrent or chronic systemic infections
* Female subjects who are pregnant, planning to become pregnant, have recently delivered, or are breast-feeding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects at Day 126 with complete closure of the PG target ulcer confirmed 2 weeks later (at Day 140) and without the need for rescue treatment | Day 126

SECONDARY OUTCOMES:
The proportions of subjects at Day 126 with a reduction in the target ulcer area of ≥ 75% or ≥ 90% from baseline. | Day 126

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Coral Gables, Florida
  - North Miami Beach, Florida
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - New York, New York
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Lubbock, Texas